CLINICAL TRIAL: NCT02303431
Title: A Phase 1, Open-Label, Single-Dose, Non-Randomized Study to Evaluate Pharmacokinetics and Pharmacodynamics of Edoxaban in Pediatric Patients
Brief Title: Phase 1 Pediatric Pharmacokinetics/Pharmacodynamics (PK/PD) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DU176b-A-U157; 2015-005732-18 (EudraCT Number)
Record Dates: First submitted 2014-10-10; First posted 2014-12-01 (Estimated); Results first posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2022-12

CONDITIONS: Deep Vein Thrombosis; Venous Thromboembolism
Keywords: Pediatric; Pharmacokinetics (PK); Pharmacodynamics (PDy); Anticoagulant; Safety
MeSH Terms: conditions — Venous Thrombosis; Venous Thromboembolism | interventions — edoxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Cohort 1a (Experimental): 12 to < 18 years of age: edoxaban low dose group
  Interventions: Drug: Edoxaban low dose
- Cohort 1b (Experimental): 12 to < 18 years of age: edoxaban high dose group
  Interventions: Drug: Edoxaban high dose
- Cohort 2a (Experimental): 6 to < 12 years of age: edoxaban low dose group
  Interventions: Drug: Edoxaban low dose
- Cohort 2b (Experimental): 6 to < 12 years of age: edoxaban high dose group
  Interventions: Drug: Edoxaban high dose
- Cohort 3a (Experimental): 2 to < 6 years of age: edoxaban low dose group
  Interventions: Drug: Edoxaban low dose
- Cohort 3b (Experimental): 2 to < 6 years of age: edoxaban high dose group
  Interventions: Drug: Edoxaban high dose
- Cohort 4a (Experimental): 6 months to <2 years of age: edoxaban low dose group
  Interventions: Drug: Edoxaban low dose
- Cohort 4b (Experimental): 6 months to <2 years of age: edoxaban high dose group
  Interventions: Drug: Edoxaban high dose
- Cohort 5a (Experimental): 0 to 6 months of age: edoxaban low dose group
  Interventions: Drug: Edoxaban low dose
- Cohort 5b (Experimental): 0 to 6 months: edoxaban high dose group
  Interventions: Drug: Edoxaban high dose

INTERVENTIONS:
Drug: Edoxaban low dose — Edoxaban low dose
  Arms: Cohort 1a; Cohort 2a; Cohort 3a; Cohort 4a; Cohort 5a
Drug: Edoxaban high dose — Edoxaban high dose
  Arms: Cohort 1b; Cohort 2b; Cohort 3b; Cohort 4b; Cohort 5b

SUMMARY:
This is the first evaluation of edoxaban in pediatric subjects. In this Phase 1 study, a single dose of edoxaban will be given to pediatric subjects who require anticoagulant therapy to see what the body does to the drug (pharmacokinetics) and what the drug does to the body (pharmacodynamics), and to compare if these effects are similar to those observed in adults.

DETAILED DESCRIPTION:
Phase 1, open-label, multiple-center study in pediatric patients from 0 to < 18 years of age. Patients will receive a single dose of edoxaban to match either the 30 mg (low dose) or the 60 mg (high dose) exposure in adults. Exact doses will be selected during the study on the basis of PK modeling of emerging data. If unanticipated exposures are observed, the target doses may be modified to best match expected exposure response relationships observed in adults.

Enrollment in the study will start with the low dose, highest age group (adolescents) and will continue from low to high dose in each age group and from higher to lower age groups. Enrollment in the next dose/age cohort will begin after 50% of the subjects have completed the previous dose/age cohort.

Age cohorts and dose groups: (6 participants each in low and high dose groups, for a total of 12 participants per age cohort)

* 12 to < 18 years of age
* 6 to <12 years of age
* 2 to <6 years of age
* 6 months to <2 years of age
* 0 to <6 months of age

ELIGIBILITY:
Inclusion Criteria:

* Is a pediatric subject requiring anticoagulant therapy
* Will abstain from the use of nonsteroidal anti-inflammatory drugs (such as ibuprofen), and other antiplatelet and anticoagulant agents (except for aspirin) from 24 hours prior to edoxaban dose until after the last PK sample is collected
* Will follow food and concomitant medication restrictions

Exclusion Criteria:

* Any major or clinically relevant unexplained bleeding during prior anticoagulant therapy
* History of abnormal bleeding or coagulation within last 6 months prior to study drug administration
* Renal function with glomerular filtration rate (GFR) less than 50% of normal for age and size
* Malabsorption disorders (e.g., cystic fibrosis or short bowel syndrome)
* Hepatic disease associated with coagulopathy leading to a clinically relevant bleeding risk, alanine transaminase (ALT) > 5 times the upper limit of normal (ULN) or total bilirubin > 2 times the ULN with direct bilirubin > 20% of the total

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2014-11-05 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (35):
- United States (12):
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of Colorado Denver, Denver, Colorado
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - University of Louisville ; Kosair Charities Pediatric Clincial Research Unit, Louisville, Kentucky
  - Duke University Medical Center (DUMC), Durham, North Carolina
  - University Hospitals Case Medical Center - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Hasbro Children's Hospital, Providence, Rhode Island
  - St. Jude Children's Research Hospital, Inc., Memphis, Tennessee
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - McMaster Children's Hospital, Hamilton, Ontario
  - Childrens Hospital of Eastern Ontario, Ottawa
- France (2):
  - Hopital Arnaud de Villeneuve, Montpellier
  - CHU Bordeaux - Hopital Haut-Leveque, Pessac
- India (3):
  - Nirmal Hospital Pvt. Ltd, Gujrāt
  - Institute of Child Health, Kolkata
  - Christian Medical College and Hospital, Ludhiāna
- Italy (3):
  - Istituto Giannina Gaslini - UOSD Emostasi e Trombosi, Genova
  - A O Universita degli Studi di Padova ; Dipartimento di Salute della Donna e del Bambino-Universita di Padova, Padua
  - Bambino Gesu Hospital, Rome
- Lebanon (2):
  - Hotel Dieu De France, Beirut
  - Hammoud Hospital University Medical Center, Saida
- Spain (5):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Araba, Vitoria-Gasteiz
- Ege University Medical Faculty - Department of Pediatric Hematology, Izmir, Turkey (Türkiye)
- United Kingdom (5):
  - Leeds General Infirmary, Leeds
  - Glenfield Hospital, Leicester
  - Guy's and St Thomas Hospital NHS Trust, London
  - Royal Brompton Hospital, London
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 66 participants who met all inclusion criteria and no exclusion criteria were enrolled in the study and received treatment at 32 clinical sites in the United States, Canada, France, India, Italy, Jordan, Lebanon, Spain, Turkey, and the United Kingdom.
Pre-assignment Details: Participants were asked to fast for at least 4 hours before dosing and for an additional 2 hours after dosing. If this was not feasible because of the participant's age or other needs, (unflavored) milk, or an equivalent substitute liquid (but not fruit juices), was allowed until 1 hour before and starting at 1 hour postdose (total volume of liquids not to exceed 240 mL).
Groups:
- Cohort 1a: 30 mg Edoxaban: Participants who were 12 to < 18 years of age and received a single-dose, oral tablet of 30 mg edoxaban.
- Cohort 1b: 60 mg Edoxaban: Participants who were 12 to < 18 years of age and received a single dose, oral tablet of 60 mg edoxaban.
- Cohort 2a: 24 mg Edoxaban: Participants who were 6 to < 12 years of age and received a single dose, oral suspension of 24 mg edoxaban.
- Cohort 2b: 45 mg Edoxaban: Participants who were 6 to < 12 years of age and received a single dose, oral suspension of 45 mg edoxaban.
- Cohort 3a: 0.7 mg/kg Edoxaban: Participants who were 2 to < 6 years of age and received a single dose, oral suspension of 0.7 mg/kg (cap 24 mg) edoxaban.
- Cohort 3b: 1.4 mg/kg Edoxaban: Participants who were 2 to < 6 years of age and received a single dose, oral suspension of 1.4 mg/kg (cap 45 mg) edoxaban.
- Cohort 4a: 0.75 mg/kg Edoxaban: Participants who were 6 months to <2 years of age and received a single dose, oral suspension of 0.75 mg/kg edoxaban.
- Cohort 4b: 1.5 mg/kg Edoxaban: Participants who were 6 months to <2 years of age and received a single dose, oral suspension of 1.5 mg/kg edoxaban.
- Cohort 5a: 0.4 mg/kg Edoxaban: Participants who were 0 to 6 months of age and received a single dose, oral suspension of 0.4 mg/kg edoxaban.
- Cohort 5b: 0.8 mg/kg Edoxaban: Participants who were 0 to 6 months of age and received a single dose, oral suspension of 0.8 mg/kg edoxaban.
Period: Overall Study
Arm/Group | Cohort 1a: 30 mg Edoxaban | Cohort 1b: 60 mg Edoxaban | Cohort 2a: 24 mg Edoxaban | Cohort 2b: 45 mg Edoxaban | Cohort 3a: 0.7 mg/kg Edoxaban | Cohort 3b: 1.4 mg/kg Edoxaban | Cohort 4a: 0.75 mg/kg Edoxaban | Cohort 4b: 1.5 mg/kg Edoxaban | Cohort 5a: 0.4 mg/kg Edoxaban | Cohort 5b: 0.8 mg/kg Edoxaban
Started | 8 | 7 | 7 | 6 | 7 | 6 | 7 | 6 | 6 | 6
Completed | 8 | 7 | 7 | 6 | 7 | 6 | 7 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed in the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1a: 30 mg Edoxaban | Cohort 1b: 60 mg Edoxaban | Cohort 2a: 24 mg Edoxaban | Cohort 2b: 45 mg Edoxaban | Cohort 3a: 0.7 mg/kg Edoxaban | Cohort 3b: 1.4 mg/kg Edoxaban | Cohort 4a: 0.75 mg/kg Edoxaban | Cohort 4b: 1.5 mg/kg Edoxaban | Cohort 5a: 0.4 mg/kg Edoxaban | Cohort 5b: 0.8 mg/kg Edoxaban | Total
Number analyzed (Participants) | 8 | 7 | 7 | 6 | 7 | 6 | 7 | 6 | 6 | 6 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 7 | 7 | 6 | 7 | 6 | 7 | 6 | 6 | 6 | 66
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.9 (1.1) | 15.3 (1.3) | 9.6 (1.1) | 9.5 (1.9) | 4.3 (1.6) | 4.3 (1.4) | 1.2 (0.5) | 1.0 (0.5) | 0.2 (0.2) | 0.3 (0.2) | 6.5 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 3 | 4 | 3 | 1 | 3 | 3 | 2 | 3 | 31
  Male | 3 | 3 | 4 | 2 | 4 | 5 | 4 | 3 | 4 | 3 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 4 | 3 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 10
  White | 7 | 6 | 5 | 5 | 5 | 3 | 2 | 5 | 2 | 3 | 43
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Parameter of Apparent Systemic Clearance (CL/F)
Description: A model-based pooled population pharmacokinetic (PK) method was used to estimate systemic clearance (CL/F). As prespecified in the protocol, arms were pooled due to sparse PK samples being collected. the median PK estimate is reported in all participants at a total of 5 blood samplings.
Time Frame: 0.25 to 1 hours, 1.5 to 3 hours, 4 to 8 hours, 9 to 14 hours, and 24 to 36 hours post-dose
Population: Pharmacokinetic parameters were assessed in the Population Pharmacokinetic (PopPK) Analysis Set. As prespecified in the study protocol, PK parameters were reported from the pooled PopPK dataset in order to support dose determination in the ongoing Phase 3 DU176b-A-U312. The current pooled PopPK dataset included participants who were newborn to <18 years of age (Cohort 1 to 5) as reported in the table.
Measure: Median (90% Confidence Interval); unit: L/h
Groups:
- All Participants: All participants included in the study (Cohorts 1a, 1b, 2a, 2b, 3a, 3b, 4a, 4b, 5a, and 5b).
Arm/Group | All Participants
Number analyzed (Participants) | 64
L/h | 42.9 [40.3 to 45.6]

2. Primary Outcome: Pharmacokinetic Parameter of Apparent Volume of Distribution (V/F)
Description: A model-based pooled population pharmacokinetic (PK) method was used to estimate apparent volume of distribution (V/F). As prespecified in the protocol, arms were pooled due to sparse PK samples being collected. the median PK estimate is reported in all participants at a total of 5 blood samplings.
Time Frame: 0.25 to 1 hours, 1.5 to 3 hours, 4 to 8 hours, 9 to 14 hours, and 24 to 36 hours post-dose
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: Liters
Arm/Group | All Participants
Number analyzed (Participants) | 64
Liters | 198 [180 to 219]

3. Secondary Outcome: Pharmacodynamic Parameter Mean Prothrombin Time (PT)
Description: Descriptive statistics were used to assess Mean Prothrombin Time (PT) by cohort at a total of 6 blood samplings.
Time Frame: Pre-dose and 0.25 to 1 hours (except for Cohorts 4a, 4b, 5a, and 5b, 0.5 to 2 hours), 1.5 to 3 hours, 4 to 8 hours, 9 to 14 hours, and 24 to 36 hours post-dose
Population: Pharmacodynamic (PD) parameters were assessed in participants with available data in the Pharmacodynamic Analysis Set. PD data were not assessed at certain timepoints due to patients not being available for the analysis (ie, indicated by rows with 0 participants at certain timepoints). In addition, standard deviation was not calculated for rows with just 1 participant in the analysis; data are reported for the timepoints in which data were collected.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cohort 1a: 30 mg Edoxaban | Cohort 1b: 60 mg Edoxaban | Cohort 2a: 24 mg Edoxaban | Cohort 2b: 45 mg Edoxaban | Cohort 3a: 0.7 mg/kg Edoxaban | Cohort 3b: 1.4 mg/kg Edoxaban | Cohort 4a: 0.75 mg/kg Edoxaban | Cohort 4b: 1.5 mg/kg Edoxaban | Cohort 5a: 0.4 mg/kg Edoxaban | Cohort 5b: 0.8 mg/kg Edoxaban
Number analyzed (Participants) | 7 | 7 | 6 | 5 | 6 | 4 | 4 | 4 | 6 | 5
seconds
  Pre-dose: 0.25 to 1 hours: number analyzed (Participants) | 6 | 7 | 4 | 4 | 5 | 4 | 4 | 4 | 6 | 5
  Pre-dose: 0.25 to 1 hours | 13.3 (1.1) | 13.5 (0.5) | 14.0 (0.4) | 13.9 (0.5) | 14.6 (1.3) | 13.7 (0.5) | 13.6 (0.7) | 13.8 (1.6) | 16.3 (4.0) | 15.3 (1.8)
  Post-dose: 0.25 to 1 hours: number analyzed (Participants) | 6 | 7 | 4 | 4 | 5 | 4 | 4 | 4 | 6 | 5
  Post-dose: 0.25 to 1 hours | 15.0 (1.8) | 17.3 (4.1) | 19.1 (3.1) | 21.3 (7.0) | 18.7 (2.0) | 22.0 (0.8) | 21.4 (2.4) | 26.5 (7.6) | 18.3 (3.0) | 21.8 (4.1)
  Pre-dose: 1.5 to 3 hours: number analyzed (Participants) | 7 | 7 | 5 | 5 | 6 | 4 | 1 | 0 | 0 | 0
  Pre-dose: 1.5 to 3 hours | 13.3 (1.0) | 13.5 (0.5) | 14.0 (0.4) | 14.9 (2.2) | 14.7 (1.3) | 13.7 (0.5) | 14.3 |  |  |
  Post-dose: 1.5 to 3 hours: number analyzed (Participants) | 7 | 7 | 5 | 5 | 6 | 4 | 1 | 0 | 0 | 0
  Post-dose: 1.5 to 3 hours | 17.6 (2.5) | 23.0 (3.8) | 26.8 (14.9) | 25.3 (5.9) | 21.0 (2.5) | 21.3 (2.3) | 20.0 |  |  |
  Pre-dose: 3.5 to 6 hours: number analyzed (Participants) | 6 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pre-dose: 3.5 to 6 hours | 13.4 (1.1) | 13.6 (0.6) | 13.4 |  |  |  |  |  |  |
  Post-dose: 3.5 to 6 hours: number analyzed (Participants) | 6 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Post-dose: 3.5 to 6 hours | 17.9 (4.6) | 20.1 (2.0) | 16.5 |  |  |  |  |  |  |
  Pre-dose: 4 to 8 hours: number analyzed (Participants) | 1 | 2 | 3 | 4 | 6 | 4 | 1 | 0 | 0 | 0
  Pre-dose: 4 to 8 hours | 12.9 | 13.4 (0.1) | 14.2 (0.2) | 13.9 (0.5) | 14.7 (1.3) | 13.7 (0.5) | 14.3 |  |  |
  Post-dose: 4 to 8 hours: number analyzed (Participants) | 1 | 2 | 3 | 4 | 6 | 4 | 1 | 0 | 0 | 0
  Post-dose: 4 to 8 hours | 15.9 | 17.5 (2.3) | 17.9 (1.3) | 18.0 (2.2) | 17.3 (0.8) | 16.1 (2.0) | 17.4 |  |  |
  Pre-dose: 6.5 to 8 hours: number analyzed (Participants) | 6 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pre-dose: 6.5 to 8 hours | 13.4 (1.1) | 13.6 (0.7) | 13.7 (0.4) |  |  |  |  |  |  |
  Post-dose: 6.5 to 8 hours: number analyzed (Participants) | 6 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Post-dose: 6.5 to 8 hours | 14.7 (1.4) | 16.7 (1.5) | 15.8 (1.1) |  |  |  |  |  |  |
  Pre-dose: 9 to 14 hours: number analyzed (Participants) | 1 | 2 | 3 | 5 | 6 | 4 | 1 | 0 | 0 | 0
  Pre-dose: 9 to 14 hours | 12.9 | 13.4 (0.1) | 14.4 (0.5) | 14.9 (2.2) | 14.7 (1.3) | 13.7 (0.5) | 14.3 |  |  |
  Post-dose: 9 to 14 hours: number analyzed (Participants) | 1 | 2 | 3 | 5 | 6 | 4 | 1 | 0 | 0 | 0
  Post-dose: 9 to 14 hours | 13.9 | 15.9 (1.6) | 15.8 (1.1) | 17.7 (5.1) | 16.1 (1.2) | 16.0 (2.5) | 16.7 |  |  |
  Pre-dose: 24 to 36 hours: number analyzed (Participants) | 6 | 7 | 6 | 4 | 6 | 4 | 1 | 0 | 0 | 0
  Pre-dose: 24 to 36 hours | 13.4 (1.1) | 13.5 (0.5) | 14.2 (0.5) | 13.9 (0.5) | 14.7 (1.3) | 13.7 (0.5) | 14.3 |  |  |
  Post-dose: 24 to 36 hours: number analyzed (Participants) | 6 | 7 | 6 | 4 | 6 | 4 | 1 | 0 | 0 | 0
  Post-dose: 24 to 36 hours | 13.1 (1.0) | 13.8 (0.7) | 14.5 (0.6) | 14.5 (0.9) | 15.5 (0.9) | 14.9 (1.1) | 14.1 |  |  |

4. Secondary Outcome: Pharmacodynamic Parameter Mean Activated Partial Thromboplastin Time (aPTT)
Description: Descriptive statistics were used to assess Mean Activated Partial Thromboplastin Time by cohort for a total of 6 blood samplings.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cohort 1a: 30 mg Edoxaban | Cohort 1b: 60 mg Edoxaban | Cohort 2a: 24 mg Edoxaban | Cohort 2b: 45 mg Edoxaban | Cohort 3a: 0.7 mg/kg Edoxaban | Cohort 3b: 1.4 mg/kg Edoxaban | Cohort 4a: 0.75 mg/kg Edoxaban | Cohort 4b: 1.5 mg/kg Edoxaban | Cohort 5a: 0.4 mg/kg Edoxaban | Cohort 5b: 0.8 mg/kg Edoxaban
Number analyzed (Participants) | 7 | 7 | 5 | 5 | 6 | 4 | 4 | 4 | 6 | 5
seconds
  Pre-dose: 0.25 to 1 hours: number analyzed (Participants) | 6 | 7 | 3 | 5 | 4 | 4 | 4 | 4 | 6 | 5
  Pre-dose: 0.25 to 1 hours | 24.1 (1.5) | 26.0 (1.6) | 33.9 (6.4) | 32.7 (2.8) | 34.3 (4.1) | 40.7 (21.0) | 32.9 (5.3) | 34.9 (8.2) | 41.0 (17.9) | 47.7 (13.0)
  Post-dose: 0.25 to 1 hours: number analyzed (Participants) | 6 | 7 | 5 | 5 | 4 | 4 | 4 | 4 | 6 | 5
  Post-dose: 0.25 to 1 hours | 26.6 (2.0) | 28.4 (4.8) | 57.9 (26.3) | 42.4 (9.9) | 39.4 (6.4) | 45.3 (20.1) | 45.4 (6.3) | 46.0 (10.9) | 39.5 (3.8) | 52.6 (18.1)
  Pre-dose: 1.5 to 3 hours: number analyzed (Participants) | 7 | 7 | 5 | 5 | 6 | 4 | 1 | 0 | 0 | 0
  Pre-dose: 1.5 to 3 hours | 24.1 (1.4) | 26.0 (1.6) | 34.6 (5.8) | 32.7 (2.8) | 30.10 (7.2) | 40.7 (21.0) | 37.4 |  |  |
  Post-dose: 1.5 to 3 hours: number analyzed (Participants) | 7 | 7 | 5 | 5 | 6 | 4 | 1 | 0 | 0 | 0
  Post-dose: 1.5 to 3 hours | 27.7 (1.1) | 32.8 (3.0) | 62.5 (35.7) | 43.0 (3.9) | 38.1 (8.9) | 45.5 (7.9) | 40.9 |  |  |
  Pre-dose: 3.5 to 6 hours: number analyzed (Participants) | 6 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pre-dose: 3.5 to 6 hours | 23.8 (1.1) | 26.1 (1.9) | 32.2 |  |  |  |  |  |  |
  Post-dose: 3.5 to 6 hours: number analyzed (Participants) | 6 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Post-dose: 3.5 to 6 hours | 26.9 (1.4) | 30.8 (1.5) | 39.0 |  |  |  |  |  |  |
  Pre-dose: 4 to 8 hours: number analyzed (Participants) | 1 | 2 | 5 | 4 | 6 | 4 | 1 | 0 | 0 | 0
  Pre-dose: 4 to 8 hours | 26.2 | 25.5 (0.7) | 33.9 (6.4) | 32.8 (3.2) | 30.1 (7.2) | 40.7 (21.0) | 37.4 |  |  |
  Post-dose: 4 to 8 hours: number analyzed (Participants) | 1 | 2 | 5 | 4 | 6 | 4 | 1 | 0 | 0 | 0
  Post-dose: 4 to 8 hours | 24.4 | 28.9 (1.0) | 35.5 (4.9) | 38.8 (5.7) | 36.7 (10.1) | 35.7 (4.6) | 35.8 |  |  |
  Pre-dose: 6.5 to 8 hours: number analyzed (Participants) | 6 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pre-dose: 6.5 to 8 hours | 23.8 (1.1) | 26.7 (1.7) | 32.2 |  |  |  |  |  |  |
  Post-dose: 6.5 to 8 hours: number analyzed (Participants) | 6 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Post-dose: 6.5 to 8 hours | 26.4 (1.2) | 30.2 (2.3) | 34.5 |  |  |  |  |  |  |
  Pre-dose: 9 to 14 hours: number analyzed (Participants) | 1 | 2 | 2 | 5 | 6 | 4 | 1 | 0 | 0 | 0
  Pre-dose: 9 to 14 hours | 26.2 | 25.5 (0.7) | 35.8 (7.6) | 32.7 (2.8) | 30.1 (7.2) | 40.7 (21.0) | 37.4 |  |  |
  Post-dose: 9 to 14 hours: number analyzed (Participants) | 1 | 2 | 2 | 5 | 6 | 4 | 1 | 0 | 0 | 0
  Post-dose: 9 to 14 hours | 23.7 | 27.7 (0.3) | 35.3 (2.8) | 35.9 (5.7) | 33.8 (7.4) | 35.1 (7.3) | 35.0 |  |  |
  Pre-dose: 24 to 36 hours: number analyzed (Participants) | 6 | 7 | 5 | 5 | 5 | 4 | 1 | 0 | 0 | 0
  Pre-dose: 24 to 36 hours | 24.4 (1.3) | 26.0 (1.6) | 32.0 (5.6) | 32.7 (2.8) | 29.9 (8.1) | 40.7 (21.0) | 37.4 |  |  |
  Post-dose: 24 to 36 hours: number analyzed (Participants) | 6 | 7 | 5 | 5 | 5 | 4 | 1 | 0 | 0 | 0
  Post-dose: 24 to 36 hours | 24.8 (0.9) | 25.8 (1.9) | 29.0 (2.2) | 38.2 (10.7) | 32.9 (5.2) | 86.1 (112.6) | 32.5 |  |  |

5. Secondary Outcome: Pharmacodynamic Parameter Mean Anti-Factor Xa (FXa)
Description: Descriptive statistics were used to assess Mean Anti-Factor Xa (FXa) by cohort for a total of 6 blood samplings.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Cohort 1a: 30 mg Edoxaban | Cohort 1b: 60 mg Edoxaban | Cohort 2a: 24 mg Edoxaban | Cohort 2b: 45 mg Edoxaban | Cohort 3a: 0.7 mg/kg Edoxaban | Cohort 3b: 1.4 mg/kg Edoxaban | Cohort 4a: 0.75 mg/kg Edoxaban | Cohort 4b: 1.5 mg/kg Edoxaban | Cohort 5a: 0.4 mg/kg Edoxaban | Cohort 5b: 0.8 mg/kg Edoxaban
Number analyzed (Participants) | 7 | 7 | 5 | 5 | 6 | 5 | 4 | 4 | 6 | 5
IU/mL
  Pre-dose: 0.25 to 1 hours: number analyzed (Participants) | 6 | 7 | 5 | 5 | 5 | 5 | 4 | 4 | 6 | 5
  Pre-dose: 0.25 to 1 hours | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.1) | 0.1 (0.0) | 0.5 (0.3) | 0.1 (0.1) | 0.4 (0.4)
  Post-dose: 0.25 to 1 hours: number analyzed (Participants) | 6 | 7 | 5 | 5 | 5 | 5 | 4 | 4 | 6 | 5
  Post-dose: 0.25 to 1 hours | 0.5 (0.4) | 1.0 (1.0) | 1.8 (0.3) | 1.6 (0.8) | 1.2 (0.6) | 1.9 (0.2) | 2.0 (0.0) | 2.0 (0.0) | 1.1 (0.8) | 1.7 (0.7)
  Pre-dose: 1.5 to 3 hours: number analyzed (Participants) | 7 | 7 | 5 | 5 | 6 | 5 | 1 | 0 | 0 | 0
  Pre-dose: 1.5 to 3 hours | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.1) | 0.1 |  |  |
  Post-dose: 1.5 to 3 hours: number analyzed (Participants) | 7 | 7 | 5 | 5 | 6 | 5 | 1 | 0 | 0 | 0
  Post-dose: 1.5 to 3 hours | 1.3 (0.4) | 2.6 (1.0) | 1.3 (0.7) | 1.9 (0.1) | 1.7 (0.3) | 1.9 (0.2) | 2.0 |  |  |
  Pre-dose: 3.5 to 6 hours: number analyzed (Participants) | 6 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pre-dose: 3.5 to 6 hours | 0.1 (0.0) | 0.1 (0.0) | 0.1 |  |  |  |  |  |  |
  Post-dose: 3.5 to 6 hours: number analyzed (Participants) | 6 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Post-dose: 3.5 to 6 hours | 0.9 (0.4) | 1.7 (0.4) | 1.4 |  |  |  |  |  |  |
  Pre-dose: 4 to 8 hours: number analyzed (Participants) | 1 | 2 | 3 | 5 | 6 | 5 | 1 | 0 | 0 | 0
  Pre-dose: 4 to 8 hours | 0.1 | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.1) | 0.1 |  |  |
  Post-dose: 4 to 8 hours: number analyzed (Participants) | 1 | 2 | 3 | 5 | 6 | 5 | 1 | 0 | 0 | 0
  Post-dose: 4 to 8 hours | 1.0 | 1.2 (0.7) | 0.8 (0.3) | 1.5 (0.3) | 0.7 (0.2) | 0.8 (0.6) | 1.2 |  |  |
  Pre-dose: 6.5 to 8 hours: number analyzed (Participants) | 6 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pre-dose: 6.5 to 8 hours | 0.1 (0.0) | 0.1 (0.0) | 0.1 |  |  |  |  |  |  |
  Post-dose: 6.5 to 8 hours: number analyzed (Participants) | 6 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Post-dose: 6.5 to 8 hours | 0.4 (0.1) | 0.9 (0.4) | 0.8 |  |  |  |  |  |  |
  Pre-dose: 9 to 14 hours: number analyzed (Participants) | 1 | 2 | 2 | 5 | 6 | 5 | 1 | 0 | 0 | 0
  Pre-dose: 9 to 14 hours | 0.1 | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.1) | 0.1 |  |  |
  Post-dose: 9 to 14 hours: number analyzed (Participants) | 1 | 2 | 2 | 5 | 6 | 5 | 1 | 0 | 0 | 0
  Post-dose: 9 to 14 hours | 0.4 | 0.6 (0.3) | 0.3 (0.1) | 0.8 (0.5) | 0.2 (0.1) | 0.4 (0.2) | 0.3 |  |  |
  Pre-dose: 24 to 36 hours: number analyzed (Participants) | 6 | 7 | 5 | 5 | 6 | 5 | 1 | 0 | 0 | 0
  Pre-dose: 24 to 36 hours | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.0) | 0.1 (0.1) | 0.1 |  |  |
  Post-dose: 24 to 36 hours: number analyzed (Participants) | 6 | 7 | 5 | 5 | 6 | 5 | 1 | 0 | 0 | 0
  Post-dose: 24 to 36 hours | 0.1 (0.0) | 0.1 (0.1) | 0.1 (0.0) | 0.2 (0.1) | 0.3 (0.5) | 0.4 (0.7) | 0.1 |  |  |

6. Other Pre Specified Outcome: Mean Palatability Score for the Liquid Formulation on a 100 mm Visual Analog Scale (VAS)
Description: Overall palatability, bitterness, sweetness, and overall taste or aroma were assessed by participants (or guardians) receiving the liquid oral suspension where each subscale used a 100 mm visual analog scale (VAS), where a 0 score corresponded to a sad face and indicated a low palatability, bitter (sharp, pungent taste or smell), not sweet, and no aroma score (eg, patients not pleased; worse outcome in terms of palatability) and a 100 score corresponded to a happy face and indicated a high palatability, not bitter, very sweet, very tasty, and high aroma score (eg, patients were pleased; best outcome in terms of palatability). Patients who were old enough scored the VAS themselves. For younger children, the parents provided this information, if possible. For the youngest children, there was free text input available to provide information on whether the patient spat it out or may not have liked the flavor, etc.
Time Frame: Baseline up to 30 minutes post-dose
Population: Palatability scores were assessed in patients who received an oral suspension of edoxaban.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Cohort 2a: 24 mg Edoxaban | Cohort 2b: 45 mg Edoxaban | Cohort 3a: 0.7 mg/kg Edoxaban | Cohort 3b: 1.4 mg/kg Edoxaban | Cohort 4a: 0.75 mg/kg Edoxaban | Cohort 4b: 1.5 mg/kg Edoxaban | Cohort 5a: 0.4 mg/kg Edoxaban | Cohort 5b: 0.8 mg/kg Edoxaban
Number analyzed (Participants) | 7 | 6 | 7 | 6 | 7 | 6 | 6 | 6
mm
  Overall palatability: number analyzed (Participants) | 7 | 6 | 7 | 6 | 6 | 6 | 6 | 6
  Overall palatability | 53.6 (35.8) | 63.2 (48.9) | 55.3 (40.6) | 83.3 (20.4) | 77.3 (27.7) | 73.0 (22.9) | 67.3 (18.4) | 83.2 (14.1)
  Bitterness: number analyzed (Participants) | 7 | 5 | 7 | 6 | 6 | 6 | 6 | 6
  Bitterness | 66.1 (44.5) | 53.2 (46.3) | 40.6 (43.5) | 66.7 (37.6) | 77.5 (27.2) | 36.3 (41.2) | 47.0 (32.6) | 65.7 (36.8)
  Sweetness: number analyzed (Participants) | 7 | 6 | 7 | 6 | 5 | 6 | 6 | 6
  Sweetness | 39.1 (34.9) | 54.3 (36.9) | 65.9 (42.1) | 81.7 (21.6) | 86.2 (26.1) | 76.2 (20.2) | 68.5 (19.0) | 86.0 (13.3)
  Overall taste: number analyzed (Participants) | 7 | 5 | 7 | 6 | 6 | 6 | 6 | 6
  Overall taste | 57.9 (42.3) | 78.2 (43.2) | 62.6 (44.9) | 83.3 (25.8) | 82.8 (24.3) | 80.5 (10.0) | 70.8 (17.0) | 85.2 (11.2)
  Aroma: number analyzed (Participants) | 7 | 6 | 7 | 6 | 6 | 6 | 6 | 6
  Aroma | 53.4 (38.4) | 57.7 (34.00) | 58.7 (39.5) | 75.0 (27.4) | 84.5 (23.9) | 72.3 (19.7) | 73.2 (13.9) | 74.2 (23.3)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected after the participant (or parent/guardian) signed the informed consent form and through the follow-up visit, up to 10 days after the single dose of exodaban.
Description: A TEAE is defined as an adverse event that emerges during treatment, having been absent pretreatment, or worsening relative to the pretreatment state.
Arm/Group | Cohort 1a: 30 mg Edoxaban | Cohort 1b: 60 mg Edoxaban | Cohort 2a: 24 mg Edoxaban | Cohort 2b: 45 mg Edoxaban | Cohort 3a: 0.7 mg/kg Edoxaban | Cohort 3b: 1.4 mg/kg Edoxaban | Cohort 4a: 0.75 mg/kg Edoxaban | Cohort 4b: 1.5 mg/kg Edoxaban | Cohort 5a: 0.4 mg/kg Edoxaban | Cohort 5b: 0.8 mg/kg Edoxaban
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/7 | 0/6 | 0/7 | 0/6 | 0/7 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7 | 0/7 | 0/6 | 0/7 | 0/6 | 0/7 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/8 | 2/7 | 4/7 | 2/6 | 1/7 | 0/6 | 3/7 | 1/6 | 0/6 | 0/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1a: 30 mg Edoxaban (N=8) | Cohort 1b: 60 mg Edoxaban (N=7) | Cohort 2a: 24 mg Edoxaban (N=7) | Cohort 2b: 45 mg Edoxaban (N=6) | Cohort 3a: 0.7 mg/kg Edoxaban (N=7) | Cohort 3b: 1.4 mg/kg Edoxaban (N=6) | Cohort 4a: 0.75 mg/kg Edoxaban (N=7) | Cohort 4b: 1.5 mg/kg Edoxaban (N=6) | Cohort 5a: 0.4 mg/kg Edoxaban (N=6) | Cohort 5b: 0.8 mg/kg Edoxaban (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT02303431/Prot_SAP_000.pdf